CLINICAL TRIAL: NCT06651723
Title: Incidence Assessment of Gingival Fissures Associated with the Use of Manual and Electric Toothbrushes: a Randomized Clinical Trial
Brief Title: Incidence Assessment of Gingival Fissures Associated with the Use of Manual and Electric Toothbrushes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Rui Vicente Oppermann, PhD, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 60844322.5.0000.5347
Record Dates: First submitted 2024-10-18; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-01

CONDITIONS: Gingival Recession; Gingival Abrasion; Wounds and Injuries
Keywords: Gingival fissures; Gingival recession; Risk factors; Traumatic toothbrushing
MeSH Terms: conditions — Gingival Recession; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The study will be blind randomized crossover clinical trial of 2 months' duration. The randomization will occur at day 0, followed by the 1st phase (30 days), a washout period of 21 days, and finally the 2nd phase (30 days).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electric brushes (Experimental): The participants will use an electric soft brush (test).
  Interventions: Device: Toothbrush type
- Manual brushes (Active Comparator): The participants will use a soft manual brush (control).
  Interventions: Device: Toothbrush type

INTERVENTIONS:
Device: Toothbrush type — The participants will use either an electric soft brush (test) and soft manual brush (control).

SUMMARY:
Gingival fissures (GF) have been suggested as risk indicators for clinical attachment loss (CAL) and gingival recession, especially in free surfaces and in patients with low plaque scores. The major factors related to the GF occurrence are high daily brushing frequencies, excessive force to brush, malpositioned teeth, use of abrasive dentifrices, and stiffness of the toothbrushes bristles. Thus, in order to better understand the pathogenesis and progression of GF, this study aim to evaluate the incidence of GF in young adults using manual and electric soft toothbrushes, in a cross-over randomized clinical trial along 2 months.

DETAILED DESCRIPTION:
Sample:

* Sample Calculation: The sample size calculation was based on the study by Greggianin et al., (2013) considering the smallest differences between means present. The result determined 28 participants in a crossover study, with a significance level of 0.05; study power of 0.8 according to calculations performed on the website: http://hedwig.mgh.harvard.edu/sample_size/js/js_crossover_quant.html. Considering an attrition rate of 20%, the number of participants included should be 34.
* Recruitment: Students duly enrolled in high school classes at Colégio Tiradentes, Porto Alegre/RS, will be invited to participate in this study. The sample will be recruited from the verbal invitation by the researchers in the classroom. The invitation will contain the study objectives, volunteer profile, inclusion and exclusion criteria, a summary of the research procedures, as well as the risks and benefits that the study will bring to the participants, and contact information for the researchers. At the end of this invitation, the students will receive the informed consent form for participants over the age of 18 or the parent/guardian informed consent form + ICF. These terms must be returned signed within one week in case of interest in participating in the study. The following week, those interested in participating who return the terms will undergo a dental examination to confirm their inclusion in the study. If eligible, they will be scheduled to begin the study.

Oral hygiene tools:

* Hand brushes: toothbrushes with soft texture, multi-strand, small head and flat surface will be purchased, by the researchers, in the local market from the same manufacturer, type and lot.
* Electric toothbrushes: electric toothbrushes will be obtained in the local market from the same manufacturer, type and lot. In this study, soft tips will be used, with a small oval head, multiple bristle, flat and soft. The electric toothbrushes have a straight, flat handle, and are waterproof.
* Toothpaste: fluoride toothpastes, with no therapeutic action, of low abrasion (containing silica) will be distributed to the participants according to their consumption. The dentifrices, belonging to the same lot, will be purchased by the researchers in the local market.

Assessment procedures:

* Interview: At the beginning of the study (day 0), an interview will be conducted, in which the participants will answer a questionnaire about their sociodemographic data and oral hygiene habits. Frequency, timing, and predominant brushing technique, as well as the type of toothbrush used and use of interdental plaque control devices will be recorded. Estimated time and reason for toothbrush change will also be recorded. At the end of the experimental phase, the volunteers will answer a questionnaire about the perceived use of the brushes provided.
* Clinical Evaluation of Gingival Fissures: A clinical examination to evaluate the presence of GF will be conducted on the buccal surfaces of all teeth, except third molars. After washing and lightly drying the teeth and gums, a staining solution (Basic Fuchsin 1%, aqueous solution) will be applied with a cotton tip. After one minute, the area will be washed with a jet of water and dried again to examine for the presence of GF. The measurement of the GF will be performed with the aid of a North Carolina periodontal probe, positioned following the path of the GF from the gingival margin to the most apical portion of the lesion. The results observed will be recorded in a specific form, prepared to register the path, extension and location of the GF that appear during the study. A trained examiner (D.G.S.) will be responsible for assessing and recording the GF. The examiner will be trained by a senior examiner (R.V.O.) and calibrated to record the presence of GF by analyzing twenty randomized images of GF photographs from the study database and repeating these analyses at a one-week interval. Agreement between assessments will be statistically tested using the Intraclass Correlation Index (ICI) and Kappa test. Before the start of the study, reproducibility values above 0.7 are expected.
* Periodontal Exam: A clinical periodontal examination will be conducted on all teeth present except third molars. Visible Plaque Index (VPI) and Gingival Bleeding Index (GBI) will be performed on buccal, lingual/palatal and proximal sites. Bleeding on Probing (BoP), Periodontal Probing Depth (PPD) and Clinical Attachment Loss (CAL) will be performed on 6 sites per tooth. PPD and CAL will be measured in millimeters and rounded up when necessary using a North Carolina type probe. Two calibrated examiners (D.G.S; M. L. B. M) will be responsible for the examinations. Calibration will be performed prior to the start of the study, the examiners will be trained to record VPI, GBI and BoP and calibrated to record the PPD and CAL exams, under the supervision of a senior researcher (RVO). Reproducibility of the PPD and CAL exams will be obtained from repeating the exams on 10 of the participants, with a minimum interval of one hour. Agreement between assessments will be statistically tested using the ICI and Kappa test. Before the beginning of the study, we expect reproducibility values above 0.7.

Data Collection:

The research consultations will be performed in the Colégio Tiradentes of the Military Brigade of Porto Alegre, with the necessary facilities and approvals. Thus, a dental office unit, bench for materials, containing toilet and dental chair, equipped with reflector, triple syringe and spittoon, will be used. The preparation of the space will follow the biosafety guidelines of the Biosafety Working Group - UFRGS.

Experimental Design

* Pre-experimental procedures: Participants will receive a dental prophylaxis with the aid of manual scaling for the removal of dental calculus and other retentive factors, polishing of tooth surfaces with prophylactic paste, rubber cup and floss 21 days before the start of the experimental phase.
* Experimental Period: At the beginning of the study (day 0, baseline), the participants will answer questionnaire 1, followed by periodontal and then GF exams. After that, the participants will be allocated to one of the two experimental groups: TG = electric brushes; CG = manual brushes, using a randomization table available at www.random.org.br. The randomization will be performed by a researcher not involved in the tests (P. D. M. A.) and the results will be stored in a sealed brown envelope. The same researcher will then distribute the corresponding oral hygiene kits. Participants will be informed to maintain their regular oral hygiene habits and instructed on how to operate the electric toothbrushes according to the manufacturer's instructions. New toothpaste will be provided as demand throughout the study upon return of the used tube. Participants will be advised not to share the toothbrush and toothpaste with people in their household. The clinical evaluation of the presence of GF will be performed at 15 and 30 days, while periodontal clinical parameters will be measured on the 30th day. At the end of the first experimental phase, the kits used will be collected by the researchers and the participants will receive a new dental prophylaxis, after which they will enter a 21-day wash out period, where they should return to their regular oral hygiene habits. At the end of this wash out period, the second experimental phase will begin. The participants will receive a new oral hygiene kit, containing the second toothbrush. The second phase of the study will follow the experimental sequence of the first phase and, at the end, they will return the oral hygiene kit, receive a new dental prophylaxis and fill out the questionnaire about the perception of the use of the two brushes. Photographs may be taken with the patient's agreement for illustrative records of the study.
* Adverse Event Reporting and Stopping Rule: Participants will be required to report, during the study, any adverse effects they may experience associated with the use of the oral hygiene kit. In case of detection of attachment loss ≥ 3 mm, treatment will be discontinued, and the participant will be followed up until remission of the GF.

ELIGIBILITY:
Inclusion Criteria:

Good systemic health (ASA I and II); No history of periodontitis (no interproximal bone loss ≥ 3 mm); No gingival recession ≥ 3 mm; Minimum number of 20 teeth.

Exclusion Criteria:

Use of medications that alter in some way the gingival and/or periodontal inflammatory response (phenytoin, sodium valproate, nifedipine, verapramil, diltiazem amlodipine, felodipine, cyclosporine [Murakami et al., 2018]); Having had antibiotic therapy in the last three months; Crowding; Presence of restorations and/or carious lesions in the cervical region on the buccal surfaces; Being under orthodontic treatment; Type 1 or 2 Diabetes Mellitus; Being a smoker; Being pregnant; Presence of full crowns and/or implants; Need for antibiotic prophylaxis for periodontal examination;

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Gingival fissures | From enrollment to the end of experimental time (2 months)
  Clinical examination, under disclosing solution, will evaluate the presence of gingival fissures (GF) on the buccal surfaces of all teeth, except third molars. Additionally, the measurement of the GF will be performed with the aid of a North Carolina periodontal probe, positioned following the path of the GF from the gingival margin to the most apical portion of the lesion.

SECONDARY OUTCOMES:
Toothbrush wear | From enrollment to the end of experimental time (2 months)
  The participants will be oriented to return the toothbrushes used at the end of each experimental phase. The toothbrush deformation/wear will be investigated by comparing the dimensions of height, width and length, in anterior, middle and posterior parts of the toothbrush (measured with a digital caliper), before and after its use by the participants, in each phase of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Rui V Oppermann, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Faculdade de Odontologia, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No